CLINICAL TRIAL: NCT00017446
Title: Phase II Evaluation Of CP4071 In Previously Treated Advanced Sarcomas
Brief Title: CP4071 in Treating Patients With Locally Advanced or Metastatic Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068689; CPMC-IRB-9825; NCI-G01-1952
Record Dates: First submitted 2001-06-06; First posted 2003-06-12 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-09

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Digitoxin

INTERVENTIONS:
Drug: CP4071

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of CP4071 in treating patients who have locally advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy, in terms of response rate, of CP4071 in patients with previously treated, locally advanced or metastatic soft tissue sarcoma.
* Determine the clinical toxic effects of this drug in these patients.

OUTLINE: Patients receive oral CP4071 daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed soft tissue sarcoma

  * Metastatic or locally advanced
  * Failed at least 1 prior therapy
* Measurable disease outside prior irradiation field
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine less than 1.5 times ULN
* Calcium less than ULN
* Potassium normal

Other:

* No other malignancy within the past 5 years except stage I or II cancer in complete remission, carcinoma in situ of the cervix, or basal cell or squamous cell skin cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic response modifier therapy allowed

Chemotherapy:

* No more than 3 prior chemotherapy regimens for advanced, recurrent, or metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy for malignancy

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior surgery and recovered

Other:

* No other concurrent cardiac glycosides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States